CLINICAL TRIAL: NCT01600183
Title: Safety and Efficacy of the Universal Neonatal Foot Orthosis in the Treatment of Metatarsus Adductus (MTA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unfo Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNFO-12-SOR-CTIL
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Metatarsus Adductus; Metatarsus Varus
Keywords: MTA; metatarsus; Metatarsus Adductus, also known as Metatarsus Varus
MeSH Terms: conditions — Metatarsus Varus | interventions — POLR1G protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- casting (Active Comparator): subjects with MTA will be treated with cast for 20 weeks. casting is replaced during every study visit.
  Interventions: Procedure: cast
- UNFO-s (Experimental): subjects with MTA will be treated with the UNFO-s device for 12 weeks - will be worn day and night during first 6 weeks and only at night during next 6 weeks
  Interventions: Device: UNFO-s

INTERVENTIONS:
Device: UNFO-s — The UNFO-s is a foot orthosis used to treat congenital foot malformations in infants
  Arms: UNFO-s
Procedure: cast — casting of the infant legs
  Arms: casting

SUMMARY:
This is a prospective, randomized, control, open label study in which up to 50 subjects with metatarsus adductus (MTA) will be enrolled. Subjects will be treated with the standard casting or using the UNFO-s device for total time of 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with an acute MTA that did not receive any treatment for this condition
* Consenting parents
* Ages 1-4 months

Exclusion Criteria:

* Participation in another clinical trial.
* Neuromuscular disorders
* Any condition which in the opinion of the investigator renders the subject ineligible for study participation.

Ages: 1 Month to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Healing of the MTA | 20 weeks
  Healing of the MTA: straightening of the foot with apprx. 10% overcorrection

SECONDARY OUTCOMES:
safety of the UNFO-s device | 7 months
  Safety is defined as absence of serious complications associated with the use of the investigational device within 2 month of the last visit.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Atar, Prof, Principal Investigator — Soroka MC
Locations (1):
- Soroka MC, Beersheba, Israel